CLINICAL TRIAL: NCT04928170
Title: The Halland Osteoarthritis (HALLOA) Cohort Study - a Five-year Observational Longitudinal Study With Focus on Metabolic Osteoarthritis
Brief Title: The Halland Osteoarthritis Cohort
Acronym: HALLOA
Status: Active, not recruiting | Type: Observational
Sponsor: FoU Center Spenshult (Other)
Collaborators: The Swedish Rheumatism Ass (Other)
Responsible Party: Sponsor
Other Study IDs: HALLOA
Record Dates: First submitted 2021-02-02; First posted 2021-06-16 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Osteoarthritis, Knee; Osteoarthritis Hand; Osteoarthritis Generalized
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and EDTA plasma
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HALLOA: 306 individuals with knee pain in the age between 30 and 65 years, without cruciate ligament injury

SUMMARY:
Osteoarthritis is the most common musculoskeletal disease and is characterized by cartilage destruction, osteophyte formation, subchondral bone sclerosis and cysts. Modern treatment strategies, as well as preventive measures, include early detection and knowledge of the early course of the disease. This includes how stress patterns, physical activity, impaired function and metabolic changes and other comorbidities affect development and possible associations with osteoarthritis.

The overall objective was to study the early development of osteoarthritis of the knee and its association with hand- and general osteoarthritis, metabolic diseases, biomarkers, long-term pain, physical function and stress patterns

DETAILED DESCRIPTION:
The overall objective was to study the early development of osteoarthritis of the knee and its association with hand- and general osteoarthritis, metabolic diseases, biomarkers, long-term pain, physical function and stress patterns.

The project includes 4 different research areas that are studied with the help of several smaller sub-studies:

Research area 1: Metabolic osteoarthritis - to study the connections between metabolic factors and osteoarthritis development in the knee and hand.

A. Relationship between knee osteoarthritis and metabolic factors B. Relationship between osteoarthritis of the hand and metabolic factors Research area 2: Biomarkers in knee and hand osteoarthritis - to study cartilage and bone markers that reflect different processes in osteoarthritis development, e.g. inflammation, matrix degradation both in the short and long term Research area 3: Pain and osteoarthritis - to study pain development and pain pressure thresholds in relation to lifestyle, depression and health-related quality of life in individuals with symptomatic knee osteoarthritis Research area 4: Physical function and osteoarthritis - to study physical function, physical activity and measured stress patterns, as well as changes in stress patterns and the relationship between these and the development of osteoarthritis over time.

Study design This is a longitudinal cohort study including 306 individuals with knee pain in the southwest of Sweden, the Halland osteoarthritis (HALLOA) cohort. The enrolments took place from 2017-2019. The participants were recruited: 1) by primary health care clinics when searching care for knee pain, or 2) by advertisements in local newspapers. The inclusion criterions were current knee pain, aged 30-65 years, with no former known radiographic knee osteoarthritis (RKOA). the exclusion criterions were no cruciate ligament rupture or rheumatologic disorder. A general practitioner examined all participants to confirm the exclusion criteria.

The cohort will be followed for five years with yearly follow-ups.

ELIGIBILITY:
Inclusion Criteria:

Knee pain

Exclusion Criteria:

Cruciate ligament injury and rheumatic disease (RA, PsoA, As, Sponylarthritis etc)

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 306 individuals with knee pain without cruciate ligament injury, age between 30 and 65 years
Sampling Method: Probability Sample
Enrollment: 312 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
BMI (kg/m2) | At baseline
  weight (kg) and height (m) are meassured and BMI will be calculated
BMI (kg/m2) | At 2 years follow-up
  weight (kg) and height (m) are meassured and BMI will be calculated
BMI (kg/m2) | At 5 years follow-up
  weight (kg) and height (m) are meassured and BMI will be calculated
Abdominal circumference (cm) | At baseline
  Abdominal circumference are meassured with measuring tape at navel height
Abdominal circumference (cm) | At 2 years follow-up
  Abdominal circumference are meassured with measuring tape at navel height
Abdominal circumference (cm) | At 5 years follow-up
  Abdominal circumference are meassured with measuring tape at navel height
Body composition | At baseline
  Body composition are assessed by Inbody 770, which gives data on proportion of muscle and body fat (separate meassures on visceral fat
Body composition | At 2 years follow-up
  Body composition are assessed by Inbody 770, which gives data on proportion of muscle and body fat (separate meassures on visceral fat
Body composition | At 5 years follow-up
  Body composition are assessed by Inbody 770, which gives data on proportion of muscle and body fat (separate meassures on visceral fat
Glucos | At Baseline
  Fasting glucos (mmol/L) meassured in serum
Glucos | At 1 year follow-up
  Fasting glucos (mmol/L) meassured in serum
Glucos | At 2 years follow-up
  Fasting glucos (mmol/L) meassured in serum
Glucos | At 3 years follow-up
  Fasting glucos (mmol/L) meassured in serum
Glucos | At 4 years follow-up
  Fasting glucos (mmol/L) meassured in serum
Glucos | At 5 years follow-up
  Fasting glucos (mmol/L) meassured in serum
HbA1c | At baseline
  HbA1c (mmol/mol) meassured in serum
HbA1c | At 1 year follow-up
  HbA1c (mmol/mol) meassured in serum
HbA1c | At 2 years follow-up
  HbA1c (mmol/mol) meassured in serum
HbA1c | At 3 years follow-up
  HbA1c (mmol/mol) meassured in serum
HbA1c | At 4 years follow-up
  HbA1c (mmol/mol) meassured in serum
HbA1c | At 5 years follow-up
  HbA1c (mmol/mol) meassured in serum
Total-cholesterol | At baseline
  Total-cholesterol (mmol/L) meassured in serum
Total-cholesterol | At 1 year follow-up
  Total-cholesterol (mmol/L) meassured in serum
Total-cholesterol | At 2 years follow-up
  Total-cholesterol (mmol/L) meassured in serum
Total-cholesterol | At 3 years follow-up
  Total-cholesterol (mmol/L) meassured in serum
Total-cholesterol | At 4 years follow-up
  Total-cholesterol (mmol/L) meassured in serum
Total-cholesterol | At 5 years follow-up
  Total-cholesterol (mmol/L) meassured in serum
Triglycerides | At baseline
  Triglycerides (mmol/L) meassured in serum
Triglycerides | At 1 year follow-up
  Triglycerides (mmol/L) meassured in serum
Triglycerides | At 2 years follow-up
  Triglycerides (mmol/L) meassured in serum
Triglycerides | At 3 years follow-up
  Triglycerides (mmol/L) meassured in serum
Triglycerides | At 4 years follow-up
  Triglycerides (mmol/L) meassured in serum
Triglycerides | At 5 years follow-up
  Triglycerides (mmol/L) meassured in serum
LDL-cholesterol | At baseline
  LDL-cholesterol (mmol/L) meassured in serum
LDL-cholesterol | At 1 year follow-up
  LDL-cholesterol (mmol/L) meassured in serum
LDL-cholesterol | At 2 years follow-up
  LDL-cholesterol (mmol/L) meassured in serum
LDL-cholesterol | At 3 years follow-up
  LDL-cholesterol (mmol/L) meassured in serum
LDL-cholesterol | At 4 years follow-up
  LDL-cholesterol (mmol/L) meassured in serum
LDL-cholesterol | At 5 years follow-up
  LDL-cholesterol (mmol/L) meassured in serum
HDL-cholesterol | At baseline
  HDL-cholesterol (mmol/L) meassured in serum
HDL-cholesterol | At 1 year follow-up
  HDL-cholesterol (mmol/L) meassured in serum
HDL-cholesterol | At 2 years follow-up
  HDL-cholesterol (mmol/L) meassured in serum
HDL-cholesterol | At 3 years follow-up
  HDL-cholesterol (mmol/L) meassured in serum
HDL-cholesterol | At 4 years follow-up
  HDL-cholesterol (mmol/L) meassured in serum
HDL-cholesterol | At 5 years follow-up
  HDL-cholesterol (mmol/L) meassured in serum
Sensitive C-Reactive Protein (CRP) | At baseline
  sensitive CRP (g/L) meassured in serum
Sensitive C-Reactive Protein (CRP) | At 1 year follow-up
  sensitive CRP (g/L) meassured in serum
Sensitive C-Reactive Protein (CRP) | At 2 years follow-up
  sensitive CRP (g/L) meassured in serum
Sensitive C-Reactive Protein (CRP) | At 3 years follow-up
  sensitive CRP (g/L) meassured in serum
Sensitive C-Reactive Protein (CRP) | At 4 years follow-up
  sensitive CRP (g/L) meassured in serum
Sensitive C-Reactive Protein (CRP) | At 5 years follow-up
  sensitive CRP (g/L) meassured in serum
Interleukin-1 (IL-1) | At baseline
  IL-1 (pg/mL) meassured in plasma with ELISA
Interleukin-1 (IL-1) | At 1 year follow-up
  IL-1 (pg/mL) meassured in plasma with ELISA
Interleukin-1 (IL-1) | At 2 years follow-up
  IL-1 (pg/mL) meassured in plasma with ELISA
Interleukin-1 (IL-1) | At 3 years follow-up
  IL-1 (pg/mL) meassured in plasma with ELISA
Interleukin-1 (IL-1) | At 4 years follow-up
  IL-1 (pg/mL) meassured in plasma with ELISA
Interleukin-1 (IL-1) | At 5 years follow-up
  IL-1 (pg/mL) meassured in plasma with ELISA
Interleukin-6 (IL-6) | At baseline
  IL-6 (pg/mL) meassured in plasma with ELISA
Interleukin-6 (IL-6) | At 1 year follow-up
  IL-6 (pg/mL) meassured in plasma with ELISA
Interleukin-6 (IL-6) | At 2 years follow-up
  IL-6 (pg/mL) meassured in plasma with ELISA
Interleukin-6 (IL-6) | At 3 years follow-up
  IL-6 (pg/mL) meassured in plasma with ELISA
Interleukin-6 (IL-6) | At 4 years follow-up
  IL-6 (pg/mL) meassured in plasma with ELISA
Interleukin-6 (IL-6) | At 5 years follow-up
  IL-6 (pg/mL) meassured in plasma with ELISA
Tumor Necrosis Factor-alfa (TNF-alfa) | At baseline
  TNF-alfa (pg/mL) meassured in plasma with ELISA
Tumor Necrosis Factor-alfa (TNF-alfa) | At 1 year follow-up
  TNF-alfa (pg/mL) meassured in plasma with ELISA
Tumor Necrosis Factor-alfa (TNF-alfa) | At 2 years follow-up
  TNF-alfa (pg/mL) meassured in plasma with ELISA
Tumor Necrosis Factor-alfa (TNF-alfa) | At 3 years folllow-up
  TNF-alfa (pg/mL) meassured in plasma with ELISA
Tumor Necrosis Factor-alfa (TNF-alfa) | At 4 years follow-up
  TNF-alfa (pg/mL) meassured in plasma with ELISA
Tumor Necrosis Factor-alfa (TNF-alfa) | At 5 years follow-up
  TNF-alfa (pg/mL) meassured in plasma with ELISA
Leptin | At baseline
  Leptin (ng/mL) meassured in serum with ELISA
Leptin | At 1 year follow-up
  Leptin (ng/mL) meassured in serum with ELISA
Leptin | At 2 years follow-up
  Leptin (ng/mL) meassured in serum with ELISA
Leptin | At 3 years follow-up
  Leptin (ng/mL) meassured in serum with ELISA
Leptin | At 4 years follow-up
  Leptin (ng/mL) meassured in serum with ELISA
Leptin | At 5 years follow-up
  Leptin (ng/mL) meassured in serum with ELISA
Galectin-1 | At baseline
  Galectin-1 (ng/mL) meassured in plasma with ELISA
Galectin-1 | At 1 year follow-up
  Galectin-1 (ng/mL) meassured in plasma with ELISA
Galectin-1 | At 2 years follow-up
  Galectin-1 (ng/mL) meassured in plasma with ELISA
Galectin-1 | At 3 years follow-up
  Galectin-1 (ng/mL) meassured in plasma with ELISA
Galectin-1 | At 4 years follow-up
  Galectin-1 (ng/mL) meassured in plasma with ELISA
Galectin-1 | At 5 years follow-up
  Galectin-1 (ng/mL) meassured in plasma with ELISA
One-leg rise | At baseline
  Knee strenght are assessed by one-leg rise
One-leg rise | At 2 years follow-up
  Knee strenght are assessed by one-leg rise
One-leg rise | At 5 years follow-up
  Knee strenght are assessed by one-leg rise
30s-chair stand test | At baseline
  Knee strenght are assessed by 30s-chair stand test
30s-chair stand test | At 2 years follow-up
  Knee strenght are assessed by 30s-chair stand test
30s-chair stand test | At 5 years follow-up
  Knee strenght are assessed by 30s-chair stand test
Maximal voluntary isometric contraction of Quadriceps | At baseline
  Maximal voluntary isometric contraction of Quadriceps assessed by dynamometer (N)
Maximal voluntary isometric contraction of Quadriceps | At 2 years follow-up
  Maximal voluntary isometric contraction of Quadriceps assessed by dynamometer (N)
Maximal voluntary isometric contraction of Quadriceps | At 5 years follow-up
  Maximal voluntary isometric contraction of Quadriceps assessed by dynamometer (N)
Hand strenght | At baseline
  Hand strenght are assessed by grippit (N)
Hand strenght | At 2 years follow-up
  Hand strenght are assessed by grippit (N)
Hand strenght | At 5 years follow-up
  Hand strenght are assessed by grippit (N)
Fitness | At 2 years follow-up
  Fitness are assessed by Åstrands test
Fitness | At 5 years follow-up
  Fitness are assessed by Åstrands test
Pain thresholds | At baseline
  pain threshold are assesed by computerized pressure algometry on eight predefined tender points out of the 18 points as part of the definition of fibromyalgia
Pain thresholds | At 2 years follow-up
  pain threshold are assesed by computerized pressure algometry on eight predefined tender points out of the 18 points as part of the definition of fibromyalgia
Pain thresholds | At 5 years follow-up
  pain threshold are assesed by computerized pressure algometry on eight predefined tender points out of the 18 points as part of the definition of fibromyalgia
Knee injury and osteoarthritis outcome score (KOOS) | At baseline
  KOOS consists of 5 subscales, assessing self reported knee pain, other Symptoms, Function in daily living (ADL), Function in sport and recreation (Sport/Rec) and knee related Quality of life (QOL).
Knee injury and osteoarthritis outcome score (KOOS) | At 1 year follow-up
  KOOS consists of 5 subscales, assessing knee pain, other Symptoms, Function in daily living (ADL), Function in sport and recreation (Sport/Rec) and knee related Quality of life (QOL).
Knee injury and osteoarthritis outcome score (KOOS) | At 2 years follow-up
  KOOS consists of 5 subscales, assessing knee pain, other Symptoms, Function in daily living (ADL), Function in sport and recreation (Sport/Rec) and knee related Quality of life (QOL).
Knee injury and osteoarthritis outcome score (KOOS) | At 3 years follow-up
  KOOS consists of 5 subscales, assessing knee pain, other Symptoms, Function in daily living (ADL), Function in sport and recreation (Sport/Rec) and knee related Quality of life (QOL).
Knee injury and osteoarthritis outcome score (KOOS) | At 4 years follow-up
  KOOS consists of 5 subscales, assessing knee pain, other Symptoms, Function in daily living (ADL), Function in sport and recreation (Sport/Rec) and knee related Quality of life (QOL).
Knee injury and osteoarthritis outcome score (KOOS) | At 5 years follow-up
  KOOS consists of 5 subscales, assessing knee pain, other Symptoms, Function in daily living (ADL), Function in sport and recreation (Sport/Rec) and knee related Quality of life (QOL).
Pain mannequin | At baseline
  Patient reported pain distribution
Pain mannequin | At 1 year follow-up
  Patient reported pain distribution
Pain mannequin | At 2 years follow-up
  Patient reported pain distribution
Pain mannequin | At 3 years follow-up
  Patient reported pain distribution
Pain mannequin | At 4 years follow-up
  Patient reported pain distribution
Pain mannequin | At 5 years follow-up
  Patient reported pain distribution
Pain intensity | At baseline
  Patient reported pain intensity by NRS scale 0-10 (best to worst)
Pain intensity | At 1 year follow-up
  Patient reported pain intensity by NRS scale 0-10 (best to worst)
Pain intensity | At 2 years follow-up
  Patient reported pain intensity by NRS scale 0-10 (best to worst)
Pain intensity | At 3 years follow-up
  Patient reported pain intensity by NRS scale 0-10 (best to worst)
Pain intensity | At 4 years follow-up
  Patient reported pain intensity by NRS scale 0-10 (best to worst)
Patient intensity | At 5 years follow-up
  Patient reported pain intensity by NRS scale 0-10 (best to worst)
Radiographic assessment of the knees | At baseline
  radiographic assessment of tibiofemoral- and patellofemoral joint in the knee
Radiographic assessment of the knees | At 1 year follow-up
  radiographic assessment of tibiofemoral- and patellofemoral joint in the knee
Radiographic assessment of the knees | At 2 years follow-up
  radiographic assessment of tibiofemoral- and patellofemoral joint in the knee
Radiographic assessment of the knees | At 3 years follow-up
  radiographic assessment of tibiofemoral- and patellofemoral joint in the knee
Radiographic assessment of the knees | At 4 years follow-up
  radiographic assessment of tibiofemoral- and patellofemoral joint in the knee
Radiographic assessment of the knees | At 5 years follow-up
  radiographic assessment of tibiofemoral- and patellofemoral joint in the knee
Radiographic assessment of the hands | At 2 years follow-up
  Radiographic assessment of the hands.
Radiographic assessment of the hands | At 5 years follow-up
  Radiographic assessment of the hands.
Mechanical load | At inclusion
  Movement behavior measured with a triaxle accelerometer at work and leisure over 7 days
Mechanical load | At 2 years follow-up
  Movement behavior measured with a triaxle accelerometer at work and leisure over 7 days
Mechanical load | At 5 years follow-up
  Movement behavior measured with a triaxle accelerometer at work and leisure over 7 days

SECONDARY OUTCOMES:
Blood samples for biobanking | At baseline
  serum and plasma for biobanking in -70 degrees celcius
Blood samples for biobanking | At 1 year follow-up
  serum and plasma for biobanking in -70 degrees celcius
Blood samples for biobanking | At 2 years follow-up
  serum and plasma for biobanking in -70 degrees celcius
Blood samples for biobanking | At 3 years follow-up
  serum and plasma for biobanking in -70 degrees celcius
Blood samples for biobanking | At 4 years follow-up
  serum and plasma for biobanking in -70 degrees celcius
Blood samples for biobanking | At 5 years follow-up
  serum and plasma for biobanking in -70 degrees celcius
Patient reported physical activity | At baseline
  Patient reported physical activity with questions duration and intensity according to WHO recommendations
Patient reported physical activity | At 1 year follow-up
  Patient reported physical activity with questions duration and intensity according to WHO recommendations
Patient reported physical activity | At 2 years follow-up
  Patient reported physical activity with questions duration and intensity according to WHO recommendations
Patient reported physical activity | At 3 years follow-up
  Patient reported physical activity with questions duration and intensity according to WHO recommendations
Patient reported physical activity | At 4 years follow-up
  Patient reported physical activity with questions duration and intensity according to WHO recommendations
Patient reported physical activity | At 5 years follow-up
  Patient reported physical activity with questions duration and intensity according to WHO recommendations
Patient reported smoking and snuff habits | At baseline
  Patient reported smoking habits, year for smoke or snuff cessation, number of cigarettes or amount of snuff
Patient reported smoking and snuff habits | At 1 years follow-up
  Patient reported smoking habits, year for smoke or snuff cessation, number of cigarettes or amount of snuff
Patient reported smoking and snuff habits | At 2 years follow-up
  Patient reported smoking habits, year for smoke or snuff cessation, number of cigarettes or amount of snuff
Patient reported smoking and snuff habits | At 3 years follow-up
  Patient reported smoking habits, year for smoke or snuff cessation, number of cigarettes or amount of snuff
Patient reported smoking and snuff habits | At 4 years follow-up
  Patient reported smoking habits, year for smoke or snuff cessation, number of cigarettes or amount of snuff
Patient reported smoking and snuff habits | At 5 years follow-up
  Patient reported smoking habits, year for smoke or snuff cessation, number of cigarettes or amount of snuff
Patient reported diets | At baseline
  Patient reported diets and intake of fruits and sweets
Patient reported diets | At 1 year follow-up
  Patient reported diets and intake of fruits and sweets
Patient reported diets | At 2 years follow-up
  Patient reported diets and intake of fruits and sweets
Patient reported diets | At 3 years follow-up
  Patient reported diets and intake of fruits and sweets
Patient reported diets | At 4 years follow-up
  Patient reported diets and intake of fruits and sweets
Patient reported diets | At 5 years follow-up
  Patient reported diets and intake of fruits and sweets
Patient reported alcohol habits | At baseline
  Patient reported alcohol habis assessed by AUDIT C
Patient reported alcohol habits | At 1 year follow-up
  Patient reported alcohol habis assessed by AUDIT C
Patient reported alcohol habits | At 2 years follow-up
  Patient reported alcohol habis assessed by AUDIT C
Patient reported alcohol habits | At 3 years follow-up
  Patient reported alcohol habis assessed by AUDIT C
Patient reported alcohol habits | At 4 years follow-up
  Patient reported alcohol habis assessed by AUDIT C
Patient reported alcohol habits | At 5 years follow-up
  Patient reported alcohol habis assessed by AUDIT C
Hospital Anxiety and Depression Scale (HADS) | At baseline
  HADS is a simple self-assessment form that shows a measure of the patient's mood.
Hospital Anxiety and Depression Scale (HADS) | At 1 year follow-up
  HADS is a simple self-assessment form that shows a measure of the patient's mood.
Hospital Anxiety and Depression Scale (HADS) | At 2 years follow-up
  HADS is a simple self-assessment form that shows a measure of the patient's mood.
Hospital Anxiety and Depression Scale (HADS) | At 3 years follow-up
  HADS is a simple self-assessment form that shows a measure of the patient's mood.
Hospital Anxiety and Depression Scale (HADS) | At 4 years follow-up
  HADS is a simple self-assessment form that shows a measure of the patient's mood.
Hospital Anxiety and Depression Scale (HADS) | At 5 years follow-up
  HADS is a simple self-assessment form that shows a measure of the patient's mood.
Health literacy | At 2 years follow-up
  Health literacy assessed with the Swedish Functional Health Literacy scale
Health literacy | At 3 years follow-up
  Health literacy assessed with the Swedish Functional Health Literacy scale
Health literacy | At 5 years follow-up
  Health literacy assessed with the Swedish Functional Health Literacy scale
Clinical examination of the knees | At baseline
  Clinical examination to assessing clinical knee OA
Clinical examination of the knees | At 2 years follow-up
  Clinical examination to assessing clinical knee OA
Clinical examination of the knees | At 5 years follow-up
  Clinical examination to assessing clinical knee OA
Clinical examination of the hands | At baseline
  Clinical examination of the hands assessing clinical hand OA
Clinical examination of the hands | At 2 years follow-up
  Clinical examination of the hands assessing clinical hand OA
Clinical examination of the hands | At 5 years follow-up
  Clinical examination of the hands assessing clinical hand OA
Blood pressure | At baseline
  Blood pressure assessed in sitting position after rest, mmHg
Blood pressure | At 2 years follow-up
  Blood pressure assessed in sitting position after rest, mmHg
Blood pressure | At 5 years follow-up
  Blood pressure assessed in sitting position after rest, mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Maria LE Andersson, ass.prof., Principal Investigator — FoU Spenshult
Locations (1):
- Spenshult Research and Development center (FoU Spenshult), Halmstad, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tornblom M, Haglund E, Bremander A, Nilsdotter A, Andersson ML, Hettiarachchi P, Johansson PJ, Svartengren M, Aili K. Associations between knee pain and knee-loading physical activities at work and leisure - a cross-sectional study based on accelerometer measurements. BMC Musculoskelet Disord. 2025 Apr 8;26(1):345. doi: 10.1186/s12891-025-08589-w. PMID 40200207
- [Derived] Brogren E, Andersson M, Westenius M, Wittrup J, Zimmerman M. Associations between hand osteoarthritis, obesity and lipid metabolism: a cross-sectional study of the Halland County Osteoarthritis (HALLOA) cohort. BMC Musculoskelet Disord. 2024 Nov 22;25(1):944. doi: 10.1186/s12891-024-08073-x. PMID 39578778
- [Derived] Tornblom M, Bremander A, Aili K, Andersson MLE, Nilsdotter A, Haglund E. Development of radiographic knee osteoarthritis and the associations to radiographic changes and baseline variables in individuals with knee pain: a 2-year longitudinal study. BMJ Open. 2024 Mar 8;14(3):e081999. doi: 10.1136/bmjopen-2023-081999. PMID 38458788
- [Derived] Andersson MLE, Thoren E, Sylwander C, Bergman S. Associations between chronic widespread pain, pressure pain thresholds, leptin, and metabolic factors in individuals with knee pain. BMC Musculoskelet Disord. 2023 Aug 9;24(1):639. doi: 10.1186/s12891-023-06773-4. PMID 37559026
- [Derived] Andersson M, Haglund E, Aili K, Bremander A, Bergman S. Associations between metabolic factors and radiographic knee osteoarthritis in early disease - a cross-sectional study of individuals with knee pain. BMC Musculoskelet Disord. 2022 Oct 28;23(1):938. doi: 10.1186/s12891-022-05881-x. PMID 36307803
- [Derived] Andersson MLE, Haglund E, Aili K, Bremander A, Bergman S. Cohort profile: the Halland osteoarthritis (HALLOA) cohort-from knee pain to osteoarthritis: a longitudinal observational study in Sweden. BMJ Open. 2022 Jul 14;12(7):e057086. doi: 10.1136/bmjopen-2021-057086. PMID 35835523
- See also: Study protocol — https://pubmed.ncbi.nlm.nih.gov/35835523/